CLINICAL TRIAL: NCT06502964
Title: Double-Blind, Placebo-Controlled Study of ALTO-101 in Patients With Schizophrenia and Cognitive Impairment
Brief Title: Study of ALTO-101 in Patients With Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTO-101-201
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Cognitive Impairment
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Each participant will receive both placebo and active study drug: 10-day administration each of placebo TDS and ALTO-101T TDS (in random order), with a 6- to 14-day washout period between conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ALTO-101 (Experimental): 10 days administration of ALTO-101T transdermal delivery system
  Interventions: Drug: ALTO-101; Device: ALTO-101 Transdermal Delivery System
- Placebo (Placebo Comparator): 10 days administration of placebo transdermal delivery system
  Interventions: Drug: Placebo; Device: Placebo Transdermal Delivery System

INTERVENTIONS:
Drug: ALTO-101 — ALTO-101 patches
  Arms: ALTO-101
Device: ALTO-101 Transdermal Delivery System — ALTO-101 transdermal delivery system
  Arms: ALTO-101
Drug: Placebo — Inactive placebo patches
  Arms: Placebo
Device: Placebo Transdermal Delivery System — Placebo transdermal delivery system
  Arms: Placebo

SUMMARY:
This is a Phase 2, double-blind, placebo-controlled, two-way crossover study to compare the efficacy of ALTO-101T versus placebo in change in electroencephalogram (EEG) cognitive processing markers and measures of cognition.

Additional goals are to assess pharmacokinetic (PK), safety, and tolerability of the recently developed ALTO-101T transdermal delivery system (TDS) formulation in a patient population.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia diagnosis for at least one year
* Cognitive impairment
* Stable doses of 1-2 antipsychotic medication(s) for at least 8 weeks at Visit 2
* Positive and Negative Syndrome Scale (PANSS) score: items P1, P3-P6 ≤ 5 and item P2 and P7 ≤ 4 during screening
* Have a body mass index (BMI) ≥ 18.0 and ≤ 37.0 kg/m2 (inclusive)
* Willing to comply with all study assessments and procedures

Exclusion Criteria:

* Evidence of unstable medical condition
* Acute psychiatric decompensation or severity of symptoms requiring psychiatric hospitalization in past 6 months
* Diagnosis of schizoaffective or bipolar affective disorder, dementia, or intellectual disability
* Current episode of major depressive disorder (MDD)
* Use of mood stabilizer, clozapine, and/or daily benzodiazepine
* Current moderate or severe substance use disorder

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Theta band activity | Treatment Period 1 - Day 6 and Day 11; Treatment Period 2 - Day 6 and Day 11
  Theta band activity after 5 and 10 days of dosing of ALTO-101T compared to placebo.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] ALTO-101T compared to placebo | Treatment Period Day 1 through study completion (an average of 36 days)
  Incidence, severity, and relatedness of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and discontinuation due to TEAEs.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Site 5038, Garden Grove, California
  - Site 5063, Los Angeles, California
  - Site 5106, Orange, California
  - Site 5035, Walnut Creek, California
  - Site 5060, Hollywood, Florida
  - Site 5015, Tampa, Florida
  - Site 5064, Snellville, Georgia
  - Site 5056, Chicago, Illinois
  - Site 5062, Gaithersburg, Maryland
  - Site 5124, Belmont, Massachusetts
  - Site 5108, New York, New York
  - Site 5077, New York, New York
  - Site 5109, New York, New York
  - Site 5126, White Plains, New York

IPD SHARING:
Plan to Share IPD: No